CLINICAL TRIAL: NCT01312688
Title: The Effect Early Goal-directed Therapy on Myocardial Dysfunction and Survival in ICU Patients With Severe Sepsis and Septic Shock: A Prospective Randomized Controlled Trial
Brief Title: Early Goal-directed Therapy and Myocardial Dysfunction
Acronym: SEPT-MD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Giora Landesberg MD, DSc, Hadassah Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0034-11-HMO-CTIL
Record Dates: First submitted 2011-03-01; First posted 2011-03-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-02

CONDITIONS: Sepsis; Septic Shock; Myocardial Dysfunction
Keywords: Early Goal Directed Hemodunamic Therapy in Sepsis
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard hemodynamic therapy (Other): Standard hemodynamic therapy currently accepted in our ICU
  Interventions: Other: Early Goal Directed Hemodynamic Therapy in Sepsis
- Early Goal Directed Hemodynamic Therapy (Experimental): Early Goal Directed Hemodynamic Therapy according to the Surviving Sepsis Campaign Guidelines
  Interventions: Other: Early Goal Directed Hemodynamic Therapy in Sepsis

INTERVENTIONS:
Other: Early Goal Directed Hemodynamic Therapy in Sepsis — Early Goal Directed Hemodynamic Therapy according to the SSC guidelines

SUMMARY:
The cardiovascular system plays a central role in the pathophysiology and prognosis of sepsis, yet the correct hemodynamic management of septic patients is still vigorously debated. Despite guidelines, the use of CVP and PAOP is seriously criticized for inaccurate prediction of fluid requirement. Recently studies showed that early goal-directed therapy (EGDT) aimed at achieving a ScvO2 of ≥70% significantly improved survival of septic shock patients, yet EGDT has not been adopted by all intensivists. The investigators have recently found using 2D echocardiography in 262 patients with severe sepsis or septic shock and treated by the conventional guidelines (without ScvO2) that diastolic dysfunction and reduced stroke volume index are strong independent predictors of mortality. In the present study the investigators intend to test the effect of EGDT on resuscitation, on long term myocardial function and left ventricular volumes and on survival in ICU patients with severe sepsis and septic shock. Patients will be randomized to EGDT (resuscitation directed by ScvO2) or standard of therapy for the first six hours after diagnosis of severe sepsis or septic shock and admission to the ICU. After six hours patients in septic shock will be further monitored with non invasive cardiac output (PiCCO, Pulsion Technologies). All patients will be followed daily by 2D & 3D transthoracic echocardiography with detailed measurements of systolic and diastolic left and right ventricular volumes and functions. Patients in the EGDT group will be compared to the control group for parameters of initial resuscitation (fluid volumes, ScvO2 achieved, inotrope use), initial values from non invasive cardiac output at six hours, interventions required from institution of non invasive cardiac output, early and long term effects on cardiac function and volumes from echo measurements, and mortality. The effectiveness of EGDT will thus be examined in the short and long terms.

DETAILED DESCRIPTION:
Design: Prospective randomized controlled trial, approved (now submitted for approval) by the Institutional Review Board. Over a period of 2 years, 300 patients with severe sepsis or septic shock will be randomized to either the currently accepted standard hemodynamic treatment in our ICU or to the standard plus goal-directed therapy according to the Rivers protocol and the SSC guidelines, i.e. including the addition of ScvO2 measurements and consequently derived treatments to achieve ScvO2 ≥70% for the first 6 hours after appearance of sepsis or septic shock in the ICU (Fig. 2).

After the first 6 hours all patients in septic shock (62% of the patients according to our preliminary data) will be monitored by continuous cardiac output monitoring. Additionally, all patients will be followed daily by transthoracic echocardiography for up 19 to 5 days (Fig 3). Since the patients themselves will not be able to sign an informed consent, the inclusion to the study will be approved by the attending physician in charge of the ICU who will also be able to decide on stopping the study protocol at any time according to his clinical judgment as to the best interest of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care unit patients with severe sepsis or septic shock, age 18 or above.

Exclusion Criteria:

* Pregnant women
* Patients with known significant valvular or coronary heart disease
* Patients with poor quality echocardiography imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 2 years
  In-ICU, In-hopsital and up to 2-years survival data will be collected and compared between the groups

SECONDARY OUTCOMES:
Myocardial dysfunction | 5 days
  Systolic and diastolic myocardial function will be measured by echocardiography daily in the first 5 days of treatment and compared between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Giora Landesberg, MD, DSc, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel